CLINICAL TRIAL: NCT06800066
Title: The Impact of Cannabidiol (CBD) Health Claims at Point-of-Sale on Consumer Perceptions and Behavior: Mini Mart Randomized Control Trial (RCT)
Brief Title: RCT-Consumer Perceptions of Cannabidiol (CBD) Health Claims
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00115825; 1R01DA051542 (NIH); 40010563 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2025-01-06; First posted 2025-01-29 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-12

CONDITIONS: Prevention
Keywords: Cannabidiol (CBD); Marketing; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Conduct an in-person randomized controlled trial with a sample of CBD current users (past 30 days use), non-current users (12 months ago or more) and susceptible non users. Participants will be randomly assigned to one of 2 conditions: 1) non CBD advertising (control condition) or 2) CBD advertising (experimental condition).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Non-CBD ads) (Active Comparator): In the control condition, the Mini-Mart will display 18 advertisements that are public service announcement (PSA) - type messages. These ads are not related to any products (CBD or non-CBD products) available in the Mini-Mart.
  Interventions: Behavioral: Purchase Behavior - (Non-CBD ads)
- Experimental Arm (CBD ads) (Experimental): In the experimental condition, the Mini-Mart will display 18 different advertisements for CBD and 1 display box for a CBD product.
  Interventions: Behavioral: Purchase Behavior - (CBD ads)

INTERVENTIONS:
Behavioral: Purchase Behavior - (Non-CBD ads) — Participants will complete 1 shopping visit and will be randomly assigned to one of 2 conditions: 1) non-CBD advertising (control condition) or 2) CBD advertising (experimental condition). Each condition will have approximately 20 advertisements. In each condition, the Participant will be asked to purchase 3 products.
  Arms: Control Arm (Non-CBD ads)
Behavioral: Purchase Behavior - (CBD ads) — Participants will complete 1 shopping visit and will be randomly assigned to one of 2 conditions: 1) non-CBD advertising (control condition) or 2) CBD advertising (experimental condition). Each condition will have approximately 20 advertisements. In each condition, the Participant will be asked to purchase 3 products.
  Arms: Experimental Arm (CBD ads)

SUMMARY:
Cannabidiol (CBD) cannot be marketed as having therapeutic benefits (without FDA's approval), be false or misleading to consumers, or convey the products are approved or endorsed by the FDA. In addition, CBD cannot be marketed as a food additive or dietary supplement since it is an active ingredient in an approved drug, Epidiolex. Despite this, CBD products have been illicitly advertised to consumers with these claims including unsubstantiated health claims that promote benefits including curing cancer and preventing Alzheimer's disease. These types of claims may be influencing consumers to use CBD. This study aims to examine the impact of CBD advertising with health claims on consumer purchase behavior.

DETAILED DESCRIPTION:
Cannabidiol (CBD) products have rapidly gained popularity, spanning the retail market with a range of products that the US Food and Drug Administration (FDA) regulates including drugs, dietary supplements, food/beverages and cosmetics. The FDA mandates that CBD cannot be marketed as having therapeutic benefits (without FDA's approval), be false or misleading to consumers, or convey the products are approved or endorsed by the FDA. In addition, CBD cannot be marketed as a food additive or dietary supplement since it is an active ingredient in an approved drug, Epidiolex. Despite this, CBD products have been unlawfully advertised to consumers with these claims including unsubstantiated health claims that promote benefits including curing cancer and preventing Alzheimer's disease and providing chronic pain relief. Furthermore, there is substantial evidence that retail advertising influences consumer perceptions and behaviors for other substances (e.g. tobacco, food), but no such evidence exists for how CBD health claims impact consumer behavior. This project focuses on informing regulatory actions for CBD by evaluating the impact of health claims on consumer purchase behavior.

Setting: Participants will complete the study at the University of North Carolina (UNC) Mini Mart in North Carolina. The store replica allows researchers to experimentally evaluate the influence of retail characteristics on consumer behavior in a controlled, real-world setting. The visit will last approximately 60 minutes.

Recruitment: Adult CBD past 30 day users, non-current users (use 12 Months ago or more), and susceptible never users, ages 18-79, will be recruited to participate. To recruit participants, flyers will be posted at public locations likely to reach potential participants, such as Young Men's Christian Association (YMCA)s, public libraries, CBD shops, the bus station, and local restaurants. In addition, email advertisements will be sent out via Craigslist and appropriate listservs. Interested prospective participants will complete a screening questionnaire to determine their eligibility. If eligible, participants will be invited enroll in the study. Approximately 480 participants will complete the study.

Informed consent: After determining eligibility, participants will be scheduled for a time to arrive at the Mini-Mart to complete the shopping task. Participants will provide electronic informed consent after they check in at the Mini-Mart and prior to starting the shopping task.

Randomization: Upon arrival at the Mini-Mart, participants will be randomly assigned to one of 2 conditions: 1) non CBD advertising (control condition) or 2) CBD advertising (experimental condition). Participants will have an equal chance of being randomized to either condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-79
* U.S. Resident
* Satisfies one of the following CBD use categories:

  1. Current CBD users (past 30 day use)
  2. Non current CBD users (use 12 Months ago or more) or susceptible never-user
* Able to read and speak English
* Able to complete a survey on a computer without help
* Willing to complete a shopping task at Mini Mart

Exclusion Criteria:

* Non-English speakers
* Younger than 18 years, or older than 79 years

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Percent of participants who purchase product | Minute 15
  The primary outcome is purchase of a CBD product. The percent of participants who purchase at least one CBD product in each group (CBD ads vs non-CBD ads) will be reported.

SECONDARY OUTCOMES:
Number of benefits of CBD | Minute 15
  Twelve items will measure participants' perceptions about the possible benefits of CBD - the mean number of selected benefits for each group (CBD ads vs non-CBD ads). Reporting the mean number of benefits selected (out of 12).
product safety scores | Minute 15
  During the post shopping task survey, the Participant will randomly view 1 (out of 11) CBD-labeled products that were available to purchase in the Mini-Mart. The participant will respond to a one-item measure that assesses the extent to which the participant perceives that the CBD product is safe to consume. Response options are on a 1 to 5 scale, with higher scores representing more perceived safety (i.e. 1- Not at all safe to 5- Extremely safe). The overall mean score and response option frequencies for all products combined for each group (CBD ads vs non-CBD ads) will be reported.
Willingness to try CBD (non-current CBD users) scores | Minute 15
  One item will be used to measure willingness to try CBD. Response items are on a 1 to 5 scale, with higher scores representing more likelihood to try CBD (i.e. 1- Extremely Unlikely to 5- Extremely Likely). The mean score and response option frequencies of each group (CBD ads vs non CBD ads) will be reported.

OTHER OUTCOMES:
Outcome scores | Minute 15
  Eleven items will measure participants' perceptions about the possible outcomes of CBD. Response items are on a 1 to 4 scale, with higher scores representing more agreement with the stated effect (i.e. 1- Strongly disagree to 4- Strongly agree). The mean score and response option frequencies of each item for each group (CBD ads vs non-CBD ads) will be reported.
Product Appeal scores | Minute 15
  During the post shopping task survey, the Participant will randomly view 1 (out of 11) CBD-labeled products that were available to purchase in the Mini-Mart. The Participant will respond to a one-item measure that assesses the extent to which the product is appealing to them. Response options are on a 1 to 5 scale, with higher scores representing more appeal (i.e. 1- Not at all appealing to 5- Extremely appealing). The overall mean score and response option frequencies for all products combined for each group (CBD ads vs non-CBD ads) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Wagoner, DrPH, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-06-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT06800066/ICF_000.pdf